CLINICAL TRIAL: NCT00011141
Title: Lactobacillus Plantarum as Therapy for NK-T Cell Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR06020-0165
Record Dates: First submitted 2001-02-12; First posted 2001-02-14 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Diabetes Mellitus
Keywords: Immune-mediated diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: Oral lactobacillus administration

SUMMARY:
The etiology of immune-mediated diabetes mellitus (IMD) remains unclear. However, previous studies indicate that autoimmunity may be a result of dysfunction of natural killer T cells (NK-T cells). Newly diagnoses patients with IMD have been shown in our laboratory to have significantly lower NK-T cells than normal controls. Other studies have shown that oral administration of lactobacillus can boost NK-T cell activity in children with HIV without side effects. Our objective is to evaluate the effect of lactobacillus administration on NK-T cell activity in patients with IMD

ELIGIBILITY:
Recently diagnosed (within the last 6 months) patients with immune-mediated (type 1) diabetes

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University, New York, New York, United States